CLINICAL TRIAL: NCT04907383
Title: Prospective Evaluation of Quality of Life in Patients With Acute Colonic Diverticular Disease: Diverticular Disease Registry DDR Trial
Brief Title: Prospective Evaluation of Quality of Life in Patients With Acute Colonic Diverticular Disease
Acronym: DDR
Status: Terminated | Type: Observational
Why Stopped: poor recruitment status
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 233-22042021
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Colonic Diverticulitis
Keywords: Diverticular disease; Acute diverticulitis; Emergency surgery; Prospective observational study
MeSH Terms: conditions — Diverticulitis, Colonic; Diverticular Diseases | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diverticular disease: All consecutive patients admitted to a Surgical Unit with a diagnosis of left-side colinic diverticulitis will be enrolled in the registry. Patients will be identified through their medical record numbers. One investigator in each center will obtain written informed consent from each patient and keep the patients updated on data collection.
  Inclusion criteria: 1) imaging-proven colonic diverticular disease 2) patient aged > 18 years old; 3) Written informed consent obtained. 4) A colonoscopy showing diverticular disease will be required during the follow-up or before surgical treatment if possible
  Interventions: Other: quality of life

INTERVENTIONS:
Other: quality of life — QoL assessment

SUMMARY:
A multicenter prospective observational study. Aim of the study is to identify the clinical parameters correlating with favorable outcomes in patients undergoing surgery or medical treatment for diverticular disease. The primary aim is be the assessment of quality of life of theses patients according to the GIQLY score at 1 year from the enrollment in the registry. Patients will be enrolled in a prospective study and followed for 36 months after the diagnosis of acute diverticulitis. All participating centres are tertiary hospitals located in Europe .

DETAILED DESCRIPTION:
All consecutive patients admitted to a Surgical Unit with a diagnosis of left-side colinic diverticulitis will be enrolled in the registry. Patients will be identified through their medical record numbers. One investigator in each center will obtain written informed consent from each patient and keep the patients updated on data collection.

Inclusion criteria: 1) imaging-proven colonic diverticular disease 2) patient aged > 18 years old; 3) Written informed consent obtained. 4) A colonoscopy showing diverticular disease will be required during the follow-up or before surgical treatment if possible Demographic and functional data will be recorded during the first surgical visit, together with a complete clinical examination. Data regarding the symptoms of presentation and quality of life will be collected and categorized. Comorbidity Index adjusted for age will be calculated for every patient, while those >70 years old will be assessed for frailty risk using the modified Frailty Index (mFI) described by Robinson et al. Relevant medications will be listed.

Setting, (emergency room vs outpatients clinic), need for admission, treatment, emergency surgery vs delayed elective surgery vs only medical management (including percutaneous drain placement) will be recorded.

Intraoperative parameters will be recorded in the registry both for emergency procedures and elective procedures, including several technical aspects such as level of inferior mesenteric artery ligtion, type of energy device used, number and type of stapler cartridge, size of circular stapler,. Use of the laparoscopy technique, conversion rate, peritoneal lavage, surgical second look will be recorded.

Histopathological examination will be recorded in terms of length of the specimen, the presence of microscopic or macroscopic abscesses, the presence of Crohn's like reaction or of lymphocyte infiltration and the eventual presence of unknown cancer.

Post-operative complications will be reported according to the Clavien-Dindo classification 15. Length of stay and post-discharge complications will be evaluated and recorded. Application of Enhanced recovery protocols will be considered only for at least 80% of the designed colo-rectal items will be satisfied.

One investigator in each center will be responsible for the follow up data. Functional follow up will be done yearly according to the GIQLY, FSFI, IIEF, ICIQ, IPSS questionnaires.

Data will be prospectively collected using a REDCAP database by the site principal investigator for each hospital. Quarterly meetings will be set between the study coordinators and the participating centers. A data manager (GP) will regularly control the quality of the data provided

ELIGIBILITY:
Inclusion Criteria:

* imaging-proven colonic diverticular disease
* patient aged > 18 years old
* Written informed consent obtained
* A colonoscopy showing diverticular disease will be required during the follow-up or before surgical treatment if possible
* Patients undergoing surgical or medical treatment will be enrolled in the registry and undergo a 36-months follow up period.

Exclusion Criteria:

* < 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to a Surgical Unit with a diagnosis of left-side colinic diverticulitis will be enrolled in the registry. Patients will be identified through their medical record numbers. One investigator in each center will obtain written informed consent from each patient and keep the patients updated on data collection.
  All patients diagnosed with left-side colonic diverticulitis who are treated in one of the participating hospitals will be asked to participate in this cohort study. The sample size will be that obtained at the end of the 5 years of recruitment. From January 2010 to December 2019, a mean number of 26 patients per year have been operated on for diverticular disease among each of the centers involved in the study. Thus, giving a total recruiting capacity of 78 patients per year, nearly 400 patients are expected to be enrolled in a 5 years' time period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Quality of Life Index (GIQLI) | 1 year
  The primary aim is the assessment of the quality of life of these patients according to the GIQLI score at 1 year from the enrollment in the study.
  The GIQLI5 is a 36-item patient reported outcomes instrument designed to assess GI-specific health-related quality of life in clinical practice and clinical trials of patients with GI disorders. It has five domains (GI symptoms, emotion, physical function, social function and medical treatment) and subscores range from 0-4 while the total score range from 0-144. Higher scores mean better GI health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrari, MD, Principal Investigator — ASST GOM Niguarda
Locations (1):
- ASST GOM Niguarda, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Origi M, Achilli P, Calini G, Costanzi A, Monteleone M, Montroni I, Maggioni D, Cocozza E, Megna S, Totis M, Tamini N, Ziccarelli A, Filippone G, Ferrari G, Crippa J, Spinelli A, Mari GM; AIMS Academy Clinical Research Network. The Diverticular Disease Registry (DDR Trial) by the Advanced International Mini-Invasive Surgery Academy Clinical Research Network: Protocol for a Multicenter, Prospective Observational Study. Int J Surg Protoc. 2021 Aug 30;25(1):194-200. doi: 10.29337/ijsp.157. eCollection 2021. PMID 34541429